CLINICAL TRIAL: NCT02568826
Title: Tolerability, Safety and Activity of IDN5243, 4 mg Bid Intramuscularly in the Treatment of Low Back Pain. A Prospective, Open Label, Single-center, Uncontrolled Study
Brief Title: Tolerability, Safety and Activity of a Muscle Relaxant Molecule IDN5243 in Patients With Low Back Pain
Acronym: IDN5243inLBP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled in the study.
Sponsor: Indena S.p.A (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XIL02/15
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Muscle relaxant
MeSH Terms: conditions — Low Back Pain; Muscle Hypotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDN 5243 (Experimental): IDN 5243 is a new 3-glycosyl-3-Odemethylthiocolchicine derivative endowed with muscle-relaxant, anti-inflammatory and analgesic activities for intramuscular administration in 4 mg/mL vials. It will be administered twice daily for 5 consecutive days with the first administration in the morning (8.00-10.00 AM) and the second in the evening (6.00-8.00 PM).
  Interventions: Drug: 3-glycosyl-3-Odemethylthiocolchicine derivative

INTERVENTIONS:
Drug: 3-glycosyl-3-Odemethylthiocolchicine derivative — IDN 5243 is a new muscle relaxant molecule. This molecule has showed significant anti-inflammatory activity by intraperitoneal route at 10 mg/kg in both carrageenan induced oedema and granuloma tests. IDN 5243 is a new 3-glycosyl-3-Odemethylthiocolchicine derivative endowed with muscle-relaxant, anti-inflammatory and analgesic activities. The primary packaging of test formulation will be a glass vial containing a solution of IDN 5243, 4 mg/ 1 mL. The secondary package will correspond to the patient's kit and will be a box containing ten (10) vials. The box label will be provided with a tear-off label.
  Other Names: IDN 5243

SUMMARY:
This is a prospective cohort study, open-label, uncontrolled proof of concept trial. The trial objective is to evaluate the analgesic tolerability, safety and activity of IDN 5243 (3-glycosyl-3-O-demethylthiocolchicine derivative)administered intramuscularly at 4 mg b.i.d. for 5 days in the morning (8.00-10.00 AM) and in the evening (6.00-8.00 PM) in subjects with Low Back Pain (LBP).

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate in a Phase 2 A study, the analgesic tolerability, safety and activity of IDN 5243 (3-glycosyl-3-O-demethylthiocolchicine derivative) administered intramuscularly at 4mg b.i.d. for 5 days in subjects with Low Back Pain (LBP).

IDN 5243 (3-glycosyl-3-O-demethylthiocolchicine derivative) is a new muscle relaxant molecule prepared by synthesis from D-xylose and 3-O-demethylthiocolchicine.

The primary outcomes of the study will be to evaluate the systemic safety (vital signs, laboratory evaluations and incidence of adverse events) of the study drug assessed by Investigator taking into consideration the change from baseline to DAY 5, the local tolerability assessed by the patient every day during the treatment period and by Investigator.

The secondary objectives of the study will be to evaluate the analgesic activity of the study drug. Analgesic activity will be evaluated with scoring spontaneous pain. In particular, the secondary outcome of the trial will be the change of the Visual Analogue Scale (VAS Scale) score (100 mm) evaluated at baseline and at DAY 5 (Visit V5). Moreover, the evaluation of secondary parameters for the analgesic activity and changes on quality of life will be assessed.

Patients will perform a total of 6 visits: 5 visits during the treatment duration (day 1 - day 5) and a Follow-up visit (day 12) will be performed after 7 days from the end of treatment (± 2 days in the event that the visit will occur on Sunday).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients,
* 18-70 years old inclusive,
* Signed Informed consent obtained prior the inclusion in the trial,
* A diagnosis of LBP equal to or greater than 50 mm on VAS with severe or moderate lumbar muscle spasm naïve or in relapsing condition,
* Patients must have a medical history, physical and neurological examinations that support a clinical diagnosis of acute LBP that is felt down to the lower leg below the knee with the onset no longer than 30 days before Visit 1,
* Patients must be appropriate candidates for treatment with study medication in the Investigator's clinical judgment,
* Patients must be able to appropriately verbalize pain characteristics and to complete all protocol required measurements/assessments without assistance,
* Patients must be medically stable on the basis of physical examination, medical history, vital signs, and clinical laboratory tests performed at screening.

Exclusion Criteria:

* LPB of non-mechanical origin such as neoplasm, infection or inflammatory chronic disorder,
* Serum creatinine level > 1.7 mg/dL or Urea > 17 mmol/l,
* Severe to mild hepatic dysfunction,
* Abnormal blood count,
* Ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients,
* History of anaphylaxis to drugs or allergic reactions in particular, history of hypersensitivity reactions (e.g. bronchospasm, rhinitis, urticaria) to drugs including to paracetamol,
* Patients with diabetic neuropathy, post-herpetic neuralgia, osteoarthritis pain, fibromyalgia,
* History of psychosis (e.g. schizophrenia or psychotic depression) or major depression (requiring treatment), diagnosis including dementia, anxiety, mental retardation; multiple sclerosis, Parkinson's Disease, Restless Legs Syndrome,
* Significant kidney or liver disease,
* History of gastrointestinal disorders,
* Blood coagulation disorders,
* Skin conditions affecting the site of application (e.g. eczema, weeping dermatitis),
* Use of paracetamol and/or NSAIDs (NonSteroidal AntiInflammatory Drugs) within 24 h before inclusion,
* Use of topical medications applied to the painful region within 2 days before the inclusion; use of opioids within 7 days before the inclusion,
* Use of corticosteroid drugs by any route of administration within 30 days before the inclusion,
* Use of myorelaxant drugs within 3 days before the inclusion,
* Pregnant or lactating women, or women of childbearing age not using a reliable method of contraception, or women of not child-bearing potential if not permanently sterilised or if not in post-menopausal status from at least two years,
* Males not to agree to use a reliable method of contraception during the study and the follow up period, if sexually active with a female of child-bearing potential,
* History of back (cervical, thoracic or lumbosacral) pain as 50% of the time in the 1 year prior to the first visit,
* History of any LBP episode, with the exception of the current acute LBP episode, within 3 months prior to the first visit that was greater than mild in pain intensity, or was associated with disability (e.g., loss of time from work, family, or activities of daily living), or necessitated the use of an opioid (narcotic) analgesic including tramadol,
* Medical history or physical examination results that suggest the acute LBP or any of the neurological symptoms or signs are caused by a serious medical condition (e.g., fever, chills, unexplained weight loss, bowel or urinary bladder dysfunction or incontinence, bilateral leg weakness, progressive weakness, paralysis),
* There is a high probability for surgical intervention for the back pain during the projected time on the study or that there will be an increase in the severity of the leg pain or deficits,
* Had either a surgical procedure involving the spine or intervertebral discs in the lower back region within 1 year prior to Visit 1 or had >1 surgical procedure(s) involving the spine or intervertebral discs in the lower back region,
* Has any painful condition that could interfere with the study assessments or with the patient's ability to differentiate the pain associated with the acute LBP episode from pain associated with another condition,
* History of epilepsy or recurrent seizures,
* Unable or unwilling to discontinue all prohibited medications at the time of randomization and during the time of their participation in the study,
* Known or suspected history of alcohol or drug abuse based on medical history, physical examination, urine drug screening, or the Investigator's clinical judgment,
* Have filed or plan to file a worker's compensation claim for any issue related to the current acute LBP episode,
* Currently involved in litigation or plan to seek legal recourse for any issue related to their acute LBP,
* Known allergies, hypersensitivity, or intolerance to the study drug or any excipients used in their manufacture,
* Had previously been enrolled in a muscle relaxant clinical study within 30 days before the inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety (vital signs, laboratory evaluations and incidence of adverse events) | From baseline to day 5
  The primary outcome of the study will be to evaluate the systemic safety (vital signs, laboratory evaluations and incidence of adverse events) of the study drug assessed by Investigator taking into consideration the change from baseline to DAY 5.
Local tolerability (4-point scale) | From baseline to day 5
  Local tolerability assessed by the patient using a 4-point scale (where 0=none, 1=mild, 2=moderate, and 3=severe) every day during the treatment period and clinically by Investigator.

SECONDARY OUTCOMES:
Analgesic activity (spontaneous pain) by Visual Analogue Scale | From baseline to day 5
  The secondary objectives of the study will be to evaluate the analgesic activity of the study drug. Analgesic activity will be evaluated with scoring spontaneous pain. In particular, the secondary outcome of the trial will be the delta of the Visual Analogue Scale (VAS Scale) score (100 mm) evaluated from baseline to day 5 (Visit V5). The 100 mm VAS score will consider a 0 mm value as NO pain, and 100 mm value as the most SEVERE pain imaginable.
Analgesic activity by Hand-To-Floor Distance (HTFD) | On day 1 and 5
  Hand-To-Floor Distance (HTFD) evaluated by Investigator on DAY 1 and 5. HTFD will be measured by the Investigators who will ask the patients to bend forward and try to touch the floor with the fingers; the remaining distance between fingers and ground ("hand-to-floor") will be measured by means of a rule (cm).
Quality of Life by SF-36 questionnaire | From baseline to day 5
  The patient will be asked to complete the questionnaire on quality of life (SF-36 questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Ferraccioli, MD, Principal Investigator — Istituto di Reumatologia Complesso Integrato Columbus - Policlinico Gemelli Roma
Locations (1):
- Istituto di Reumatologia Complesso Integrato Columbus - Policlinico A. Gemelli, Rome, RM, Italy

REFERENCES:
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Medications for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):505-14. doi: 10.7326/0003-4819-147-7-200710020-00008. PMID 17909211
- [Background] Mellinghoff H. [Modern muscle relaxants and their clinical application]. Anaesthesist. 1994 Apr;43(4):270-82. doi: 10.1007/s001010050058. German. PMID 8179178
- [Background] Bernstein E, Carey TS, Garrett JM. The use of muscle relaxant medications in acute low back pain. Spine (Phila Pa 1976). 2004 Jun 15;29(12):1346-51. doi: 10.1097/01.brs.0000128258.49781.74. PMID 15187636
- [Background] Dillon C, Paulose-Ram R, Hirsch R, Gu Q. Skeletal muscle relaxant use in the United States: data from the Third National Health and Nutrition Examination Survey (NHANES III). Spine (Phila Pa 1976). 2004 Apr 15;29(8):892-6. doi: 10.1097/00007632-200404150-00014. PMID 15082991
- [Background] Malanga GA, Dennis RL. Use of medications in the treatment of acute low back pain. Clin Occup Environ Med. 2006;5(3):643-53, vii. doi: 10.1016/j.coem.2006.03.002. PMID 16963380
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] Wenig CM, Schmidt CO, Kohlmann T, Schweikert B. Costs of back pain in Germany. Eur J Pain. 2009 Mar;13(3):280-6. doi: 10.1016/j.ejpain.2008.04.005. Epub 2008 Jun 3. PMID 18524652
- [Background] Gore M, Sadosky A, Stacey BR, Tai KS, Leslie D. The burden of chronic low back pain: clinical comorbidities, treatment patterns, and health care costs in usual care settings. Spine (Phila Pa 1976). 2012 May 15;37(11):E668-77. doi: 10.1097/BRS.0b013e318241e5de. PMID 22146287
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Carta M, Murru L, Botta P, Talani G, Sechi G, De Riu P, Sanna E, Biggio G. The muscle relaxant thiocolchicoside is an antagonist of GABAA receptor function in the central nervous system. Neuropharmacology. 2006 Sep;51(4):805-15. doi: 10.1016/j.neuropharm.2006.05.023. Epub 2006 Jun 30. PMID 16806306